CLINICAL TRIAL: NCT03284801
Title: Management of Acute Disseminated Encephalomyelitis in Neurology Unit of Assiut University Children Hospital
Brief Title: Management Of Acute Disseminating Encephalomyelitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Alsaid Ahmed, Principle Investigator, Assiut University
Other Study IDs: ADEM
Record Dates: First submitted 2017-09-08; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Acute Disseminated Encephalomyelitis
MeSH Terms: conditions — Encephalomyelitis, Acute Disseminated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: management of acute disseminating encephalomyelitis — clinical audit on management of acute disseminating encephalomyelitis

SUMMARY:
Acute disseminated encephalomyelitis is an immune-mediated inflammatory demyelinating disease of the central nervous system, which is typically transitory and self-limiting. It is characterized by an acute or subacute encephalopathy with neurological deficits, and magnetic resonance imaging evidence of widespread demyelination that predominantly involves the white matter of the brain and spinal cord. In the absence of specific biological markers, the diagnosis of Acute disseminated encephalomyelitis is still based upon a combination of clinical and neuro imaging features and exclusion of diseases that mimic Acute disseminated encephalomyelitis

DETAILED DESCRIPTION:
Acute disseminated encephalomyelitis can occur at any age, but usually affects children and young adults. The mean age of clinical presentation in pediatric cohorts ranges from 5 to 8 years. The annual incidence of Acute disseminated encephalomyelitis is reported to be 0.4-0.8 per 100,000 and the disease more commonly affects children and young adults, probably related to the high frequency of exanthematous and other infections and vaccination in this age group.Initial symptoms and signs of Acute disseminated encephalomyelitis usually begin within 2 days to 4 weeks after a viral infection or vaccination, and include a rapid onset encephalopathy (behavioral change or altered consciousness) associated with a combination of multifocal neurological deficits, leading to hospitalization within a week. Typically Acute disseminated encephalomyelitis presents with systemic symptoms such as fever, malaise, headache, nausea, and vomiting, which may occur shortly before the appearance of neurological signs and symptoms. The clinical course is rapidly progressive, developing maximum deficits within a few days (mean 4.5 days) . A wide variety of neurological deficits have been described in pediatric patients with Acute disseminated encephalomyelitis, including: obtundation and depressed consciousness (invariable); unilateral or bilateral long tract signs (60-95%); acute hemiplegia (76%); ataxia (18-59%); meningismus (26-31%); seizures (13-35%); spinal cord involvement (24%); visual involvement (7-23%); and speech impairment or aphasia (5-21%). Cerebellar mutism and prolonged focal motor seizures in the context of Acute disseminated encephalomyelitis have been mainly reported in children younger than 5 years of age.Acute combined peripheral nervous system demyelination is not rare in children with Acute disseminated encephalomyelitis whereas it is more frequently described in adult patients, with a reported frequency of 44% in one study. A particular Acute disseminated encephalomyelitis phenotype affecting young children has been reported in association with group A beta hemolytic streptococcal infection. Prominent behavioral disturbances, dystonic movements, and basal ganglia abnormalities on MRI (in addition to typical white matter lesions) characterize this syndrome.

Supportive care in the acute stage is critical and early antiviral treatment with acyclovir (30 mg/kg/ day) is highly recommended on admission, considering that viral encephalitis and particularly herpes simplex encephalitis is the usual primary diagnosis in a child with fever, encephalopathy, seizures, and focal neurological signs. The treatment for Acute disseminated encephalomyelitis includes primarily the management of acute attacks. Corticosteroid treatment at high doses is the most widely reported therapy. Most authors recommend a brief (3-5 days) high-dose intravenous steroid course, usually methylprednisolone given at 20-30 mg/kg/day to a maximum dose of 1 g/day, or dexamethasone given at 1 mg/kg/day, followed by oral prednisone taper for 4-6 weeks . Reported treatment approaches show a wide variety in the specific steroid formulation employed, as well as in the dosing, routes of administration, and tapering regimens. Treatment with corticosteroids requires careful monitoring of blood pressure, urine glucose, and serum potassium, and administration of gastric protection. The use of immunoglobulin has been reported in several case studies either alone or in combination with corticosteroids. The recommended total dose of immunoglobulin is 2 g/kg, administered over 2-5 days. The usefulness of immunoglobulin has been reported both as a second-line treatment in steroid-unresponsive Acute disseminated encephalomyelitis cases and in patients showing recurrent or steroid-dependent demyelination.

The use of plasma exchange has been recently established as possibly effective and it may be considered as escalation therapy for steroid-unresponsive acute fulminant demyelinating diseases including Acute disseminated encephalomyelitis, multiple sclerosis, and transverse myelitis, . Plasmapheresis should be started as soon as the treatment failure is recognized. The use of this procedure in Acute disseminated encephalomyelitis has been reported in only a small number of severe cases. A median number of seven exchanges (range 2 to 20) were reported in one study. Moderate to severe anemia, symptomatic hypotension, hypocalcemia, potential transfusion reactions or transmission of transfusion-related diseases, and heparin-associated thrombocytopenia have been described in relation to therapeutic plasma exchange. There is also a risk of catheter-related complications, including thrombosis, septic infections or pneumothorax.

Acute hemorrhagic leukoencephalitis is often considered the most acute and severe form of Acute disseminated encephalomyelitis, with a universally fatal course within hours to days after the onset of neurological symptoms without treatment. Survival in pediatric patients has been reported with combined therapy including high-dose intravenous corticosteroid, immunoglobulin, Therapeutic plasma exchange, and decompressive craniotomies. Aggressive treatment strategies such as surgical decompression have to be considered and performed in patients with fulminant variants of Acute disseminated encephalomyelitis, with evidence of continued clinical deterioration due to increased intracranial pressure, unresponsive to conventional medical treatment and critical care measures.

ELIGIBILITY:
Inclusion Criteria:

* All patient presented with manifestation of acute disseminating encephalomyelitis admitted in Assiut University Children Hospital

Exclusion Criteria:

* Patients presented with viral encephalitis,bacterial meningitis
* Cases not fulfilling MRI criteria for diagnosis of acute disseminated encephalomyelitis

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - All patient presented with manifestation of acute disseminating encephalomyelitis admitted in Assiut University Children Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
clinical audit on management of acute disseminating encephalomyelitis | within one year
  To improve diagnosis and management of acute disseminated encephalomyelitis in Neurology Unit of Assiut University Children Hospital and to decrease the mortality and residual deficits from this disease.
  The aim of this audit is to measure the current practice within the Neurology Unit of Assiut University Children Hospital team in the diagnosis and management of acute disseminated encephalomyelitis against the recommendations in American Academy of Neurology guidance by using checklist and designed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Alsaid Ahmed, resident doctor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wingerchuk DM. Postinfectious encephalomyelitis. Curr Neurol Neurosci Rep. 2003 May;3(3):256-64. doi: 10.1007/s11910-003-0086-x. PMID 12691631
- [Background] Tenembaum S, Chitnis T, Ness J, Hahn JS; International Pediatric MS Study Group. Acute disseminated encephalomyelitis. Neurology. 2007 Apr 17;68(16 Suppl 2):S23-36. doi: 10.1212/01.wnl.0000259404.51352.7f. PMID 17438235
- [Background] Menge T, Kieseier BC, Nessler S, Hemmer B, Hartung HP, Stuve O. Acute disseminated encephalomyelitis: an acute hit against the brain. Curr Opin Neurol. 2007 Jun;20(3):247-54. doi: 10.1097/WCO.0b013e3280f31b45. PMID 17495616
- [Background] Dale RC, de Sousa C, Chong WK, Cox TC, Harding B, Neville BG. Acute disseminated encephalomyelitis, multiphasic disseminated encephalomyelitis and multiple sclerosis in children. Brain. 2000 Dec;123 Pt 12:2407-22. doi: 10.1093/brain/123.12.2407. PMID 11099444
- [Background] Hynson JL, Kornberg AJ, Coleman LT, Shield L, Harvey AS, Kean MJ. Clinical and neuroradiologic features of acute disseminated encephalomyelitis in children. Neurology. 2001 May 22;56(10):1308-12. doi: 10.1212/wnl.56.10.1308. PMID 11376179
- [Background] Anlar B, Basaran C, Kose G, Guven A, Haspolat S, Yakut A, Serdaroglu A, Senbil N, Tan H, Karaagaoglu E, Karli Oguz K. Acute disseminated encephalomyelitis in children: outcome and prognosis. Neuropediatrics. 2003 Aug;34(4):194-9. doi: 10.1055/s-2003-42208. PMID 12973660
- [Background] Pohl D, Tenembaum S. Treatment of acute disseminated encephalomyelitis. Curr Treat Options Neurol. 2012 Jun;14(3):264-75. doi: 10.1007/s11940-012-0170-0. PMID 22476745
- [Background] Cortese I, Chaudhry V, So YT, Cantor F, Cornblath DR, Rae-Grant A. Evidence-based guideline update: Plasmapheresis in neurologic disorders [RETIRED]: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2011 Jan 18;76(3):294-300. doi: 10.1212/WNL.0b013e318207b1f6. PMID 21242498
- [Background] Keegan M, Pineda AA, McClelland RL, Darby CH, Rodriguez M, Weinshenker BG. Plasma exchange for severe attacks of CNS demyelination: predictors of response. Neurology. 2002 Jan 8;58(1):143-6. doi: 10.1212/wnl.58.1.143. PMID 11781423